CLINICAL TRIAL: NCT00802256
Title: Comparative Evaluation of Pulpotomized Primary Molars With Mineralized Trioxide Aggregate & New Endodonthic Cement
Brief Title: Comparative Evaluation of Pulpotomized Primary Molars With Mineral Trioxide Aggregate and New Endodonthic Cement
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Iranian center for endodontic research (Unknown)
Responsible Party: Fatemeh Shekarchi, Shaheed Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 63sh138
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Pulpotomy Treatment
Keywords: pulpotomy; primary molar teeth; MTA; NEC; CEM; Primary Molar Teeth Which Require Pulpotomy Treatment
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): teeth which are treated with Mineral Trioxide Aggregate (MTA) material
  Interventions: Procedure: pulpotomy
- B (Experimental): teeth which are treated with new Endodontic Cement (NEC) material
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: pulpotomy — removal of caries and cronal pulp tissue and then restoring of tooth

SUMMARY:
A new Endodontic Cement (NEC) is being compared with mineral trioxide aggregate in pulpotomy of primary molars.

DETAILED DESCRIPTION:
Forty patient are selected randomly. Each patient has at least 2 teeth which require pulpotomy treatment. After removing of carious teeth by a low speed round bur and pulp exposure, roof of pulp chamber is removed completely by a high speed 008 fissure bur. Life tissues of pulp are removed by sharp excavator and rinsing with normal salin. Hemostat is achieved and cavity will be cleaned by 0.5% hypo chlorate solution. MTA or NEC material is mixed according to manufacturer instruction and will be placed in pulp chamber and over pulpal canal orifices for at least 1 mm. The light cure glass inomor is also mixed according to manufacturer instruction and is places over the A or B material and cured for 40 minutes. The treated tooth will be restored with a stainless steel crown or amalgam filling material.

ELIGIBILITY:
Inclusion Criteria:

* Vital pulp exposure of teeth with caries or trauma
* No clinical signs & symptoms like pain,inflammation
* No radiographic signs & symptoms like: internal resorption,external resorption, furcation involvement,pulp canal obliteration.
* The restorable tooth
* No dental treatment contraindication

Exclusion Criteria:

* Systemic diseases
* Existence of pain,inflammation or sinus tract
* No patient compliance

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Clinical features and radiographic examination | 6 monthes and one year

CONTACTS AND LOCATIONS:
Overall Officials: Fatemeh Shekarchi, student, Principal Investigator — Saheed Behesti University for Medical sciences
Locations (1):
- Saheed Behesti University for Medical sciences, Tehran, Iran